CLINICAL TRIAL: NCT02717039
Title: Pharmacogenomics of Heparin-Induced Thrombocytopenia
Acronym: PHIT
Status: Recruiting | Type: Observational
Sponsor: University of Arizona (Other)
Collaborators: American College of Clinical Pharmacy (Other)
Responsible Party: Principal Investigator, Jason H Karnes, Assistant Professor, University of Arizona
Other Study IDs: 1512277980
Record Dates: First submitted 2016-03-17; First posted 2016-03-23 (Estimated); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Heparin-induced Thrombocytopenia
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood will be stored in freezers at minus 80 degrees
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Blood Draw: A one time blood draw of 50mL or 15mL will be performed using a vein in the participants arm. Existing venous access will be used for the blood draw in preference of new venipuncture. Participants will be enrolled in equal numbers from three categories determined by their observed clinical course: (1) participants without HIT testing negative for heparin/PF4 antibodies (controls); (2) participants without HIT testing positive for heparin/PF4 antibodies (seroconversion cases); (3) participants with HIT testing positive for both heparin/PF4 antibodies (HIT cases).
  Interventions: Procedure: Blood Draw

INTERVENTIONS:
Procedure: Blood Draw — A one time blood draw of 150 milliliters will be performed using a vein in the participants arm. Existing venous access will be used for the blood draw in preference of new venipuncture.

SUMMARY:
The purpose of this research is to identify genomic markers that can predict heparin-induced thrombocytopenia (HIT), which is a very serious side effect to heparin. Heparin is commonly used to prevent blood clots and the investigators may be able to identify genomic markers which can be used to prevent heparin use in people who will get HIT.

DETAILED DESCRIPTION:
Inclusion Criteria: 18 years of age or older; Participants with heparin/PF4 antibody and SRA testing for HIT, including:

participants with negative heparin/PF4 antibodies and negative SRA (controls), participants with positive heparin/PF4 antibodies and negative SRA(seroconversion cases), participants with positive heparin/PF4 antibodies and positive SRA (HIT cases); Treatment with unfractionated heparin or low molecular weight heparin (enoxaparin, dalteparin, tinzaparin) within 7 days of blood draw Exclusion Criteria: Less than 18 years of age; Inability to give informed consent There is no randomization involved in this study. Participants will be enrolled in equal numbers from three categories: (1) participants without HIT testing negative for heparin/PF4 antibodies (controls); (2) participants without HIT testing positive for heparin/PF4 antibodies (seroconversion cases); (3) participants with HIT testing positive for both heparin/PF4 antibodies (HIT cases).

Recruitment will be facilitated through collaborators in the Coagulation Laboratory and through key study personnel in the Banner Univerisyt Medical Center - Tucson. Patients with positive and negative heparin/PF4 antibody and serotonin release assay results will be identified in the Coagulation Laboratory and the patient's provider will be approached about potential participation in research studies. If the potential participant is interested, they will be approached by study personnel for study description and possible consent. Alternatively, clinical collaborators who are consulted and participating directly in a patients care may contact a potential participant directly for willingness to participate in the study.

Patients consenting to the study will be asked to provide a one blood sample of approximately 150 milliliters. Peripheral blood mononuclear cells (PBMCs) will be isolated from this sample and stored at -80C before use in proposed experiments. Genomic DNA will also be isolated from the sample to perform HLA sequencing.

HIT will be confirmed with a functional serotonin release assay and HIT likelihood based on clinical course. Detailed data will be collected regarding participant's hospitalization, heparin dose and duration, platelet counts, surgical history, and co-morbidities. After consent of participants, a peripheral blood sample will be acquired, CD positive T cells sorted using flow cytometry, and genomic DNA isolated as previously described.

The TCR repertoire and the proportion of specific TCR variants for a particular sample will be determined using a combination of novel technologies available in the investigator's laboratory and core facilities. The TCR repertoire of a sample will be determined using next-generation sequencing technology. The new Adaptive Technologies ImmunoSEQ TCR kit is likely to be utilized as this kit has been optimized to obtain an unbiased quantitative profile of rearranged TCR alleles from a genomic DNA sample. Currently this kit is in the beta test phase and VANTAGE is one of the test sites.

TCR sequencing will be performed using multiplex PCR system to amplify rearranged TCRbeta DNA using primers specific to a functional TCR Vbeta segment as previously described. Genomic templates will be amplified and observed relative abundance of Vbeta 5.1 family TCR clonotypes will be inferred from sequence data using an expectation maximization algorithm. CDR3 motifs as defined by the international ImMunoGeneTics information system (IMGT) will be predicted based on DNA sequences. For every read, best sequence alignment against reference sequences will be computed and reads with low quality scores will be discarded. To exclude unspecific T cells due to sorting impurities and/or stimulation background, antigen-specific clones with frequencies below 1 percent will be neglected.

TCR alleles known to be important in specific DHS will be targeted using droplet digital PCR (ddPCR). The ddPCR is a new technology that provides absolute quantification (real-time PCR provides relative quantification) of target template based on oil-emulsion droplet PCR reactions. The investigator's laboratory has experience with this new technology and assays for a number of important TCR alleles have already been optimized on the ddPCR in the investigator's laboratory.

To minimize risk extra blood will be collected for this study at the same time as primary care labs are drawn whenever possible. Participants will be asked to provide 150ml of blood in order to test qualitative immune responses. The risks associated with participating in this study relate to uncommon complications of venipuncture and could include discomfort, bruising, infection, and/or blood clot formation. Patients will be monitored for safety and comfort by trained clinical personnel.

Subjects will be monitored during the course of the study for any adverse events. Serious adverse events will be reported to the IRB within 10 days of the PI's notification of the event. Non-serious adverse events or instances of noncompliance with the protocol will be reported at the time of continuing review. The trial will be monitored in an ongoing fashion. There is no DSMB nor are any interim analyses planned.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Ability to give informed consent
* Have undergone testing for heparin/PF4 antibody with or without SRA testing for HIT
* Have received treatment with unfractionated heparin or low molecular weight heparin (enoxaparin, dalteparin, tinzaparin) prior to antibody or SRA testing

Exclusion Criteria:

* Less than 18 years of age
* Pregnancy
* Hemoglobin less than 9 mg/dL (for larger 5 ounce blood draw)
* Known Human Immunodeficiency Virus (HIV) infection
* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from a hospital setting and identified based on laboratory testing for heparin-induced thrombocytopenia.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2016-03 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Serotonin Release Assay | 0-30 days
  Functional assay confirming presence of heparin-induced thrombocytopenia
Heparin/platelet factor 4 antibody | 0-30 days
  ELISA for confirming presence of heparin/PF4 antibodies necessary for HIT

CONTACTS AND LOCATIONS:
Locations (1):
- Banner University Medical Center - Tucson, Tucson, Arizona, United States